CLINICAL TRIAL: NCT05545904
Title: A Pilot Study to Evaluate the Feasibility & Acceptability of a Peer-mentor Delivered Substance Use Screening and Brief Intervention for Adolescents in Kenya
Brief Title: Feasibility of Peer-mentor Delivered Substance Use Brief Intervention for Adolescents in Kenya
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moi University (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MoiU6
Record Dates: First submitted 2022-09-11; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Following enrollment and baseline assessment, participants will be randomized to one of the two study groups (allocation ratio: 1:1) - SBI intervention or the control condition (an education session on harms of substance use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants randomized to the intervention arm will undergo a substance use screening and brief intervention delivered by the peer-mentors. Screening will be performed using the ASSIST-Y (28). The brief intervention will be delivered in a single session (20-30 minutes) using the FRAMES model i.e.(i) providing feedback on screening results (ii) ensuring responsibility on the part of the adolescents (iii) giving clear advice to stop/cut down (iv) giving menu of options (alternative healthy behaviors to engage in) (v) expressing empathy, and (vi) encouraging self-efficacy (15). The BI will be delivered for the highest scoring substance or the one the adolescent identifies as the most problematic.
  Interventions: Behavioral: Substance use brief intervention (BI)
- Control arm (Placebo Comparator): Participants assigned to the control arm will participate in a substance use education intervention. This intervention will entail review of material in the NACADA substance use education manual for adolescents, and will be followed by a question and answer session. The manual contains summarized and simple information on the harms and myths related to alcohol, tobacco, cannabis, prescription medication and khat use, substances. This education intervention will be delivered over a single 20-30 minute session by a counselor stationed at Rafiki clinic.
  Interventions: Behavioral: substance use education intervention

INTERVENTIONS:
Behavioral: Substance use brief intervention (BI) — The BI will be delivered in a single session (20-30 minutes) using motivational interviewing techniques and the FRAMES model i.e.(i) providing feedback on screening results (ii) ensuring responsibility on the part of the adolescents (iii) giving clear advice to stop/cut down (iv) giving menu of options (alternative healthy behaviors to engage in) (v) expressing empathy, and (vi) encouraging self-efficacy (15). The BI will be delivered for the highest scoring substance or the one the adolescent identifies as the most problematic.
  Arms: Intervention arm
Behavioral: substance use education intervention — This intervention will entail review of material in the NACADA substance use education manual for adolescents, and will be followed by a question and answer session. The manual contains summarized and simple information on the harms and myths related to alcohol, tobacco, cannabis, prescription medication and khat use, substances. This education intervention will be delivered over a single 20-30 minute session by a counselor stationed at Rafiki clinic.
  Arms: Control arm

SUMMARY:
Adolescent substance use is prevalent in Kenya and in the US, and is associated with significant negative health and social outcomes. Unfortunately adolescents in both regions have limited access to substance use treatment because services are costly and scarce. The aim of this study is to pilot study procedures and obtain data on intervention acceptability, fidelity and preliminary efficacy, to determine the feasibility of a definitive randomized controlled trial (RCT) of the efficacy of a peer-delivered substance use brief intervention among adolescents attending an out-patient clinic in Kenya.

DETAILED DESCRIPTION:
Background: Adolescent substance use is prevalent in Kenya and in the US, and is associated with significant negative health and social outcomes. Unfortunately adolescents in both regions have limited access to substance use treatment because services are costly and scarce. Substance use screening and brief Intervention (SBI) delivered in primary health care by peer-mentors, represents a promising strategy for overcoming these barriers to substance use treatment for adolescents.

Objective: The aim of this study is to pilot study procedures and obtain data on intervention acceptability, fidelity and preliminary efficacy, to determine the feasibility of a definitive randomized controlled trial (RCT) of the efficacy of a peer-delivered substance use SBI among adolescents attending an out-patient clinic in Kenya.

Design: The study will use both qualitative and quantitative methods to meet its objectives

Intervention: SBI includes a single session of screening using the Alcohol, Smoking & Substance Use Involvement Screening Test for Youth questionnaire (ASSIST-Y), followed by a brief intervention (20-30 minutes of motivational interviewing) for those with moderate and high risk substance use. Three peers will be trained for five days on how to deliver the SBI. The peer-mentors will receive regular supervision throughout the study implementation process.

Outcomes: SBI feasibility will be defined by the extent to which fidelity to the SBI is maintained and the preliminary effects of the SBI on substance use and quality of life outcomes. SBI acceptability will be evaluated from the perspective of the adolescents using qualitative interviews guided by Sekhon's theoretical framework of acceptability. Feasibility of conducting a future full-scale RCT will be explored by measuring outcomes such as study participation rate, willingness to be randomized, study completion rates and ability to measure effectiveness outcomes.

Investigating team and future plans: This study will be conducted by a team including faculty from Moi Teaching and Referral Hospital, faculty from Indiana University, and a team from the National Authority for Campaign Against Alcohol and drug abuse (NACADA). Our team has experience implementing and scaling peer-led substance use SBIs for adolescent populations. If the SBI and its delivery are found to be feasible and acceptable the plan is to partner with the government to conduct a full-scale multi-site RCT in Kenya and Indiana.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adolescents attending the Rafiki clinic, aged 15-24 years and who have moderate or high risk substance use as defined by the Alcohol, Smoking & Substance Use Involvement Screening Test for Youth questionnaire (ASSIST-Y) scores

Exclusion Criteria:

* The following youth will be excluded: (i) those ill during the appointment (ii) those who decline to assent/consent (iii) those already enrolled in the Fogarty project.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in substance use scores (measured using ASSIST-Y) | Change from baseline to 3 months post-intervention.
  The researchers will compare the changes in the mean ASSIST-Y scores between the two intervention and control arms

SECONDARY OUTCOMES:
Change in quality of life scores (measured using the Brief Version WHO-Quality of life tool) | Change from baseline to 3 months post-intervention.
  The researchers will compare the changes in the mean WHO-QOL scores between the intervention and control arms
Fidelity to the intervention assessed using a researcher designed rating scale | until completion of participant recruitment and follow-up, an average of 3 months
  Fidelity checklists will be developed based on key elements of the intervention. Items will be rated by the SBI trainers on a 3-point scale.
Study Participation Rate | until completion of participant recruitment and follow-up, an average of 3 months
  Number of participants who consent to take part in the study divided by the number of eligible patients. The researchers will also document reasons for refusal to participate in the study. Benchmark to establish feasibility for conducting a full-scale randomized trial: 80% of those who eligibility meet criteria consent to participate
Proportion of participants meeting inclusion criteria who get excluded | until completion of participant recruitment and follow-up, an average of 3 months
  Number of participants excluded divided by number meeting inclusion criteria. The researchers will document reasons for exclusion; Benchmark to establish feasibility for conducting a full-scale randomized trial: 80% of those meeting inclusion criteria are not excluded
Proportion of participants willing to be randomized | until completion of participant recruitment and follow-up, an average of 3 months
  Number of participants consenting to participate divided by number willing to be randomized to either study arm; Benchmark to establish feasibility for conducting a full-scale randomized trial: 80% of those consenting are willing to be randomized to either study arm
Study Completion Rate | Baseline, month 3
  Number of participants who complete both the baseline and month 3 assessments/intervention divided by the number of participants enrolled in each study arm; Benchmark to establish feasibility for conducting a full-scale randomized trial: 80% complete both baseline and month 3 assessments
Participant Burden | Baseline, month 3
  Time required to complete data collection at each assessment time point. Benchmark to establish feasibility for conducting a full-scale randomized trial: 80% of participants complete study assessments and the SBI in less than 90 minutes at baseline; and study assessments in less than 60 minutes at month 3
Data Completeness | Baseline, month 3
  Percentage of questionnaires/study measures completed; Benchmark to establish feasibility for conducting a full-scale randomized trial: 80% of those who enroll will complete at least 80% of study questionnaires/measures

CONTACTS AND LOCATIONS:
Overall Officials: FLORENCE M, JAGUGA, MMED, Principal Investigator — MOI TEACHING & REFERRAL HOSPITAL
Locations (1):
- Florence Jaguga, Eldoret, RIFT Valley, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Degenhardt L, Stockings E, Patton G, Hall WD, Lynskey M. The increasing global health priority of substance use in young people. Lancet Psychiatry. 2016 Mar;3(3):251-64. doi: 10.1016/S2215-0366(15)00508-8. Epub 2016 Feb 18. PMID 26905480
- [Background] National Institute of Drug Abuse. Principles of Adolescent Substance Use Disorder Treatment: A Research-Based Guide: Introduction | NIDA [Internet]. [cited 2022 Feb 27]. Available from: https://nida.nih.gov/publications/principles-adolescent-substance-use-disorder-treatment-research-based-guide/introduction
- [Background] Heradstveit O, Skogen JC, Hetland J, Hysing M. Alcohol and Illicit Drug Use Are Important Factors for School-Related Problems among Adolescents. Front Psychol. 2017 Jun 20;8:1023. doi: 10.3389/fpsyg.2017.01023. eCollection 2017. PMID 28676779
- [Background] Ritchwood TD, Ford H, DeCoster J, Sutton M, Lochman JE. Risky Sexual Behavior and Substance Use among Adolescents: A Meta-analysis. Child Youth Serv Rev. 2015 May;52:74-88. doi: 10.1016/j.childyouth.2015.03.005. PMID 25825550
- [Background] Gaitho D, Kumar M, Wamalwa D, Wambua GN, Nduati R. Understanding mental health difficulties and associated psychosocial outcomes in adolescents in the HIV clinic at Kenyatta National Hospital, Kenya. Ann Gen Psychiatry. 2018 Jul 10;17:29. doi: 10.1186/s12991-018-0200-8. eCollection 2018. PMID 30002721
- [Background] Lisdahl KM, Gilbart ER, Wright NE, Shollenbarger S. Dare to delay? The impacts of adolescent alcohol and marijuana use onset on cognition, brain structure, and function. Front Psychiatry. 2013 Jul 1;4:53. doi: 10.3389/fpsyt.2013.00053. eCollection 2013. PMID 23847550
- [Background] Erskine HE, Moffitt TE, Copeland WE, Costello EJ, Ferrari AJ, Patton G, Degenhardt L, Vos T, Whiteford HA, Scott JG. A heavy burden on young minds: the global burden of mental and substance use disorders in children and youth. Psychol Med. 2015 May;45(7):1551-63. doi: 10.1017/S0033291714002888. Epub 2014 Dec 23. PMID 25534496
- [Background] Richmond-Rakerd LS, Slutske WS, Wood PK. Age of initiation and substance use progression: A multivariate latent growth analysis. Psychol Addict Behav. 2017 Sep;31(6):664-675. doi: 10.1037/adb0000304. Epub 2017 Aug 14. PMID 28805408
- [Background] Zewdu S, Hanlon C, Fekadu A, Medhin G, Teferra S. Treatment gap, help-seeking, stigma and magnitude of alcohol use disorder in rural Ethiopia. Subst Abuse Treat Prev Policy. 2019 Jan 18;14(1):4. doi: 10.1186/s13011-019-0192-7. PMID 30658659
- [Background] Jaguga F, Kwobah E. A review of the public sector substance use disorder treatment and prevention systems in Kenya. Subst Abuse Treat Prev Policy. 2020 Jul 20;15(1):47. doi: 10.1186/s13011-020-00291-5. PMID 32690036
- [Background] Hoeft TJ, Fortney JC, Patel V, Unutzer J. Task-Sharing Approaches to Improve Mental Health Care in Rural and Other Low-Resource Settings: A Systematic Review. J Rural Health. 2018 Dec;34(1):48-62. doi: 10.1111/jrh.12229. Epub 2017 Jan 13. PMID 28084667
- [Background] World Health Organisation. Brief Intervention. A Manual For Use In A Manual For Use In A Manual For Use In A Manual For Use In Primary Care Primary. 2003.
- [Background] United Nations Office on drugs and Crime. International standards on drug use prevention - second updated edition [Internet]. 2018. 58 p. Available from: http://www.unodc.org/documents/prevention/standards_180412.pdf
- [Background] Harris SK, Csemy L, Sherritt L, Starostova O, Van Hook S, Johnson J, Boulter S, Brooks T, Carey P, Kossack R, Kulig JW, Van Vranken N, Knight JR. Computer-facilitated substance use screening and brief advice for teens in primary care: an international trial. Pediatrics. 2012 Jun;129(6):1072-82. doi: 10.1542/peds.2011-1624. Epub 2012 May 7. PMID 22566420
- [Background] Winters KC, Lee S, Botzet A, Fahnhorst T, Nicholson A. One-year outcomes and mediators of a brief intervention for drug abusing adolescents. Psychol Addict Behav. 2014 Jun;28(2):464-474. doi: 10.1037/a0035041. PMID 24955669
- [Background] Carney T, Johnson K, Carrico A, Myers B. Acceptability and feasibility of a brief substance use intervention for adolescents in Cape Town, South Africa: A pilot study. Int J Psychol. 2020 Dec;55(6):1016-1025. doi: 10.1002/ijop.12668. Epub 2020 Apr 13. PMID 32285449
- [Background] Peltzer K, Matseke G, Azwihangwisi M. Evaluation of alcohol screening and brief intervention in routine practice of primary care nurses in Vhembe district, South Africa. Croat Med J. 2008 Jun;49(3):392-401. doi: 10.3325/cmj.2008.3.392. PMID 18581618
- [Background] Winn LAP, Paquette KL, Donegan LRW, Wilkey CM, Ferreira KN. Enhancing adolescent SBIRT with a peer-delivered intervention: An implementation study. J Subst Abuse Treat. 2019 Aug;103:14-22. doi: 10.1016/j.jsat.2019.05.009. Epub 2019 May 14. PMID 31229188
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Humeniuk R, Ali R, Babor TF, Farrell M, Formigoni ML, Jittiwutikarn J, de Lacerda RB, Ling W, Marsden J, Monteiro M, Nhiwatiwa S, Pal H, Poznyak V, Simon S. Validation of the Alcohol, Smoking And Substance Involvement Screening Test (ASSIST). Addiction. 2008 Jun;103(6):1039-47. doi: 10.1111/j.1360-0443.2007.02114.x. Epub 2008 Mar 28. PMID 18373724
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Osborn TL, Venturo-Conerly KE, Wasil AR, Schleider JL, Weisz JR. Depression and Anxiety Symptoms, Social Support, and Demographic Factors Among Kenyan High School Students. J Child Fam Stud [Internet]. 2020 May 1 [cited 2020 Oct 22];29(5):1432-43. Available from: https://link.springer.com/article/10.1007/s10826-019-01646-8
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Musyoka CM, Mbwayo A, Donovan D, Mathai M. Alcohol and substance use among first-year students at the University of Nairobi, Kenya: Prevalence and patterns. PLoS One. 2020 Aug 28;15(8):e0238170. doi: 10.1371/journal.pone.0238170. eCollection 2020. PMID 32857791
- [Background] Gamarel KE, Brown L, Kahler CW, Fernandez MI, Bruce D, Nichols S; Adolescent Medicine Trials Network for HIV/AIDS Intervention. Prevalence and correlates of substance use among youth living with HIV in clinical settings. Drug Alcohol Depend. 2016 Dec 1;169:11-18. doi: 10.1016/j.drugalcdep.2016.10.002. Epub 2016 Oct 11. PMID 27750182
- [Background] Atwoli L, Mungla PA, Ndung'u MN, Kinoti KC, Ogot EM. Prevalence of substance use among college students in Eldoret, western Kenya. BMC Psychiatry. 2011 Feb 28;11:34. doi: 10.1186/1471-244X-11-34. PMID 21356035
- [Background] Hogue A, Henderson CE, Ozechowski TJ, Robbins MS. Evidence base on outpatient behavioral treatments for adolescent substance use: updates and recommendations 2007-2013. J Clin Child Adolesc Psychol. 2014;43(5):695-720. doi: 10.1080/15374416.2014.915550. Epub 2014 Jun 13. PMID 24926870
- [Background] Hogue A, Henderson CE, Becker SJ, Knight DK. Evidence Base on Outpatient Behavioral Treatments for Adolescent Substance Use, 2014-2017: Outcomes, Treatment Delivery, and Promising Horizons. J Clin Child Adolesc Psychol. 2018 Jul-Aug;47(4):499-526. doi: 10.1080/15374416.2018.1466307. Epub 2018 Jun 12. PMID 29893607
- [Background] World Health Organization (WHO). Optimal Mix of Health Services. 2007; Available from: https://www.who.int/mental_health/policy/services/2_Optimal Mix of Services_Infosheet.pdf
- [Background] Aalsma MC, Dir AL, Zapolski TCB, Hulvershorn LA, Monahan PO, Saldana L, Adams ZW. Implementing risk stratification to the treatment of adolescent substance use among youth involved in the juvenile justice system: protocol of a hybrid type I trial. Addict Sci Clin Pract. 2019 Sep 6;14(1):36. doi: 10.1186/s13722-019-0161-5. PMID 31492186
- [Background] Aalsma MC, Aarons GA, Adams ZW, Alton MD, Boustani M, Dir AL, Embi PJ, Grannis S, Hulvershorn LA, Huntsinger D, Lewis CC, Monahan P, Saldana L, Schwartz K, Simon KI, Terry N, Wiehe SE, Zapolski TCB. Alliances to disseminate addiction prevention and treatment (ADAPT): A statewide learning health system to reduce substance use among justice-involved youth in rural communities. J Subst Abuse Treat. 2021 Sep;128:108368. doi: 10.1016/j.jsat.2021.108368. Epub 2021 Mar 16. PMID 33867210
- [Background] Skevington SM, Dehner S, Gillison FB, McGrath EJ, Lovell CR. How appropriate is the WHOQOL-BREF for assessing the quality of life of adolescents? Psychol Health. 2014;29(3):297-317. doi: 10.1080/08870446.2013.845668. Epub 2013 Nov 6. PMID 24192254
- [Derived] Jaguga F, Aalsma MC, Enane LA, Turissini M, Kwobah EK, Apondi E, Barasa J, Kosgei G, Olando Y, Ott MA. A qualitative pilot study exploring the acceptability of a peer provider delivered substance use brief intervention from the perspective of youth in Kenya. Subst Abuse Treat Prev Policy. 2025 Feb 11;20(1):6. doi: 10.1186/s13011-025-00639-9. PMID 39934864